CLINICAL TRIAL: NCT05797025
Title: Investigation of Pressure Pain Threshold and Pinch Grip Strength in Individuals With and Without Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 83116987-761
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain
Keywords: Pressure Pain Threshold; Neck; Neck Pain; Pinch Grip Strength; Quality of life
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with neck pain (Other): To assess pressure pain threshold and pinch grip strengths.
  Interventions: Other: To assess pressure pain threshold and pinch grip strengths.
- Healthy group (Other): To assess pressure pain threshold and pinch grip strengths.
  Interventions: Other: To assess pressure pain threshold and pinch grip strengths.

INTERVENTIONS:
Other: To assess pressure pain threshold and pinch grip strengths. — To assess pressure pain threshold and pinch grip strengths.

SUMMARY:
This study aims to determine whether there is a difference in pressure pain threshold and pinch grip strength in individuals with and without chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is a common musculoskeletal disease. In chronic pain clinics, neck pain ranks second in frequency after low back pain. Lifetime prevalence is higher in workers. 51-80% of workers experience at least one episode of neck and arm pain. Neck pain symptoms may disappear spontaneously within a few weeks, while 30% of them continue as chronic neck pain. Today, studies are planned with the theory that pathology leads to deficiencies, deficiencies lead to functional limitations, and functional limitations lead to disability. Chronic neck pain increases the cost of treatment and reduces work capacity. In addition, neck pain in industrial workplaces causes loss of work days as much as low back pain. The aim of this study is to determine whether there is a difference in pressure pain threshold and pinch grip strength in individuals with and without chronic neck pain. In addition, it is aimed to examine the relationship of these parameters with quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of neck pain for more than three months,
* With any chronic disease diagnosed,
* No past or present mental illness,
* Individuals who can speak, read and write Turkish.

Exclusion Criteria:

* Having any neurological, psychiatric or cognitive disorder,
* Individuals who cannot speak, read or write Turkish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | 1 day
  Pressure pain threshold will be measured using Baseline® dolorimeter (Fabrication Enterprises, White Plains, NY, USA). Pressure pain thresholds of the upper trapezius, sternocleidomastoid, levator scapula, and suboccipital region muscles (semispinalis capitis and splenius capitis) will be evaluated. Two measurements will be taken from all muscles in the same order and with five minutes intervals. The average of the measurements will be recorded in kilograms/centimeter2 (kg/cm2). The procedure will be explained to individuals by showing them by manual palpation before testing begins. Pressure pain threshold measurement with algometer has been reported as a valid and reliable method.
Pinch grip strength | 1 day
  Baseline® pinch meter (Mechanical Pinch Gauges, NexGen Ergonomics, Inc. Montreal, Canada) will be used to assess pinch grip strength. While measuring pinch grip strength, patients will be asked to place the pinch meter between the pulp of the thumb and index finger and squeeze with all their strength. All measurements will be performed in 3 repetitions with one-minute intervals on the right and left hands. The average of the obtained values will be recorded in kilogram force.
Neck disorders | 1 day
  Neck disorders will be assessed with the Bournemouth Questionnaire (BQ). BQ consists of 7 questions that examine pain intensity, activities of daily living, social activities, anxiety, emotional aspects of depression, kinesiophobia, and ability to control pain. The items in the questionnaire are specific to patients with neck pain, and each question evaluates a different parameter. A high score indicates a high degree of discomfort. The Turkish version of the BQ has been proven to be valid and reliable.
Arm, shoulder, and hand problems | 1 day
  Arm, shoulder, and hand problems will be evaluated with the Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH). The questionnaire consists of a disability/symptom scale (11 items) and two optional scales: work (four items) and sports/performing arts (four items). In the disability/symptom scale, each item questions the severity of pain, activity-related pain, tingling, weakness and stiffness, difficulty in performing physical activity due to upper extremity problems, and the effect of upper extremity problems on social activities, work, and sleep. Answers are given on a scale of one to five, and each question is scored from 1 to 5. Scores on the three subscales of the DASH disability/symptom scale, the work scale, and the sports/performing arts scale all range from 0 (no disability) to 100 (most severe disability). The Turkish version of DASH has been reported to be valid and reliable.
General quality of life assessed by NHP | 1 day
  The Nottingham Health Profile (NHP) is a general quality of life questionnaire that measures a person's perceived health problems and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items. Questions are answered as 'yes' or 'no'. The questionnaire assesses six parameters related to health status. These parameters are; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items), and emotional reactions (9 items). Each sub-parameter is scored between 0-100. 0 indicates best health, and 100 indicates worst health. The total NHP score is derived from the sum of the subscores.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)